CLINICAL TRIAL: NCT01071005
Title: Randomized Clinical Trial of the Pharmacodynamics of Lorelin Depot 3.75Mg (Leuprorelin Acetate) Produced by Laboratório Químico Farmacêutico Bergamo LTDA. Compared to Lupron Depot ® 3.75 Mg Produced by Abbott in Healthy Subjects
Brief Title: Pharmacodynamics of Lorelin Depot (Leuprorelin Acetate - Bergamo) Compared to Lupron Depot ® (Leuprorelin Acetate - Abbot)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Azidus Brasil (Industry)
Responsible Party: Alexandre Frederico, LAL Clinica Pesquisa e Desenvolvimento Ltda
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LEUBER0409; Versão 03 - Emenda 1
Record Dates: First submitted 2009-06-04; First posted 2010-02-18 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Healthy
Keywords: Decrease serum levels of luteinizing hormone, FSH and Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (Experimental): Lorelin Depot - Bergamo
  Interventions: Drug: Lorelin Depot Bergamo
- comparator (Active Comparator): Lupron Depot® - Abbott
  Interventions: Drug: Lupron Depot - Abbott

INTERVENTIONS:
Drug: Lorelin Depot Bergamo — Lorelin Depot Bergamo, 3,75 mg, single dose.
  Arms: Test
Drug: Lupron Depot - Abbott — Lupron Depot 3,75 mg, single dose.
  Arms: comparator

SUMMARY:
The primary objective of this study is to examine, in healthy subjects, the comparative pharmacodynamics of Lorelin Depot (leuprorelin), manufactured by the Chemical Pharmaceutical Laboratory Bergamo Ltda with the product Lupron Depot ® (leuprorelin), manufactured by Abbott Laboratories Ltd, through the strength of biological markers follicle stimulating hormone (FSH), luteinizing hormone (LH) and total testosterone, associated with the activity of the substance.

Secondarily be observed safety (tolerability) of subjects in clinical research through the comparison of clinical and laboratory parameters pre-and post-study, and incidence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Accept the Informed Consent.
2. Subjects of research males aged 40 to 45 years;
3. Subject of research with body mass index greater than or equal to 19 and less than or equal to 30;
4. Be considered healthy, from the analysis of the clinical history and medical examination;
5. Laboratory tests with results outside the values considered normal, but not considered clinically relevant.

Exclusion Criteria:

1. Have donated or lost 450 mL or more of blood in the three months preceding the study;
2. Have participated in any experimental study or have taken any experimental drug in the last three months prior to the start of the study;
3. Have made regular use of medication in the last 4 weeks prior to the start of the study or have made use of any medication a week before the study began;
4. Have been hospitalized for any reason, up to 8 weeks before the study;
5. Provide history of alcohol abuse, drugs or medications, or have ingested alcohol within 48 hours prior to the period of hospitalization;
6. Have a history of liver disease, renal, pulmonary, gastrointestinal, hematological or psychiatric;
7. Amendments pressure of any etiology requiring pharmacological treatment;
8. Present history of myocardial infarction, angina and / or heart failure.

Ages: 40 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2010-08; Primary Completion 2010-10 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Decrease of serum levels of luteinizing hormone, Testosterone and FSH | 56 days

SECONDARY OUTCOMES:
Evaluation of safety through the adverse affects investigation | 56 days

CONTACTS AND LOCATIONS:
Locations (1):
- Lal Clinica Pesquisa E Desenvolvimento Ltda, Valinhos, São Paulo, Brazil